CLINICAL TRIAL: NCT04277858
Title: Phase II Study: Induction Chemotherapy Followed by Transoral Robotic Surgery and Neck Dissection for Definitive Management of Oropharyngeal Squamous Cell Carcinoma. (NECTORS Trial)
Brief Title: Neoadjuvant Chemotherapy and Transoral Robotic Surgery for Oropharyngeal Cancer.
Acronym: NECTORS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Nader Sadeghi (Other)
Collaborators: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Sponsor-Investigator, Nader Sadeghi, Professor, McGill University Health Centre/Research Institute of the McGill University Health Centre
Organization: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MP-37-2018-3443
Record Dates: First submitted 2019-12-11; First posted 2020-02-20 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Oropharynx Cancer; Tonsil Cancer; Throat Cancer; Base of the Tongue Carcinoma
Keywords: oropharynx cancer; throat cancer; HPV related throat cancer; tonsil cancer; base of tongue cancer
MeSH Terms: conditions — Oropharyngeal Neoplasms; Tonsillar Neoplasms | interventions — Docetaxel; Cisplatin

STUDY DESIGN:
Intervention Model Description: neoadjuvant Docetaxel and Cisplatin and transoral surgery
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Neoadjuvant chemotherapy and surgery (Experimental): Docetaxel and Cisplatin x 3 cycles followed by Transoral robotic surgery and neck dissection.
  Carboplatin may be used instead of Cisplatin.
  Interventions: Drug: Docetaxel

INTERVENTIONS:
Drug: Docetaxel — Subjects will be treated with neoadjuvant docetaxel and cisplatin for 3 cycles. This is followed by transoral robotic surgery (TORS) and neck dissection as definitive treatment, reserving radiotherapy for salvage.
  Other Names: Cisplatin, Transoral robotic surgery

SUMMARY:
The objective of this trial is to study the efficacy of treatment of human papilloma virus (HPV) related oropharyngeal cancer with chemotherapy followed by Transoral Robotic Surgery (TORS) as definitive treatment. Current treatment of oropharyngeal cancer are chemo-radiotherapy. There is significant lifelong side effects associated with this approach related to tissue effects of radiotherapy. The side effects results in significant quality of life deterioration among the patients. Overall there is 20% failure rate with this treatment approach. The study hypothesis is that treatment with upfront (neoadjuvant) chemotherapy followed by transoral surgery and neck dissection is highly effective treatment allowing competitive cure rate compared to chemo-radiotherapy with less than 10% failure rate, while avoiding radiotherapy in majority of cases. It is also hypothesized that better functional and quality of life outcome maybe achieved with this approach.

DETAILED DESCRIPTION:
The current standard of care for advanced (AJCC-7 edition stage III and IV) oropharyngeal squamous cell carcinoma are concomitant chemoradiation, or surgery followed by adjuvant radiation therapy with or without concomitant chemotherapy. These approaches have persistent and significant lifelong side effects and sequelae related to treatment, and in particular related to radiotherapy. The side effects of radiotherapy (augmented with concomitant chemotherapy) include soft tissue fibrosis, loss of salivary function, dry mouth, life long disturbed taste function, poor dental health with rapidly decaying teeth, dysfunction of swallowing, significant loss of the mobility of the base of tongue and pharyngeal constrictors, loss of laryngeal elevation, esophageal stricture, and at times severe side effects such as soft tissue necrosis or osteoradionecrosis of the mandible. About 10% of the patients undergoing chemoradiation for oropharyngeal cancer develop long term swallowing dysfunction with feeding tube dependency. As a result , patient's quality of life (QOL) is adversely affected. Improvements in the side effect profile of treatment, the functional outcome, and the QOL remain very important areas of advancement in treating this patient population. Improvements in functional outcome need to be achieved while maintaining or improving the oncologic outcome and cure rates for cancer, compared to the standard of care.

Use of Taxane based chemotherapy along with Platinum drugs (Cisplatin and Carboplatin) in high dose neoadjuvant setting, coupled with Transoral Laser Microsurgery (TLM) or Transoral Robotic Assisted Surgery (TORS), allows potential for improved oncologic outcome as well as avoidance of long term sequelae of high dose radiation therapy to head and neck. These transoral surgical approaches (TLM and TORS) provide improved functional outcome compared with traditional open composite resections and complex reconstructive algorithms for oropharynx. TLM and TORS are currently in clinical use for early (stage T1 and T2 with N0 or N+ve) oropharyngeal cancer.

De-escalation treatment strategies of TORS followed by adjuvant radiotherapy are being investigated currently. However even without de-escalation there is overall 18-20% rate of treatment failure and half of failures are due to distant metastasis in the absence of loco-regional recurrence. In this study the investigators propose systemic escalation of treatment with neoadjuvant chemotherapy (docetaxel and cisplatin) followed by de-escalated locoregional treatment with transoral surgery and neck dissection reserving radiotherapy for salvage.

This approach has the potential for improved functional outcome by avoiding short and more importantly long term and permanent sequelae of radiation therapy in oropharyngeal cancer treatment. This approach is a new paradigm in treatment of oropharyngeal cancer, and can significantly improve the functional outcome of cancer treatment.

ELIGIBILITY:
Inclusion Criteria:

* Squamous cell cancer of oropharynx, p 16 positive
* American Joint Commission on Cancer version-7 (AJCC-7) Stage III (T1N1, T2N1, T3N0, T3N1) and stage IVa (T1N2, T2N2, T3N2)
* Treatment Naive
* No evidence of distant metastatic disease
* Fit for surgery, and primary tumor assessed surgically resectable with negative margins via transoral approach
* Age > 18 years
* Karnofsky performance status > 60% or Eastern Cooperative Oncology Group (ECOG) < 2
* Absolute neutrophil count (ANC) > 2,000, platelets > 100,000 and calculated creatinine clearance > 50 cc/min
* Signed study specific consent form
* No other malignancies except cutaneous basal cell carcinoma (BCC) or squamous cell carcinoma (SCC) within the last 5 years
* Agree to use effective contraception while on the study. Women of child bearing potential must have a negative pregnancy test, and not be lactating.

Exclusion Criteria:

* Patients with advanced T4 cancer unresectable without organ preservation
* P16 negative tumor
* N3 disease (Stage IVB AJCC-7)
* 5 or more positive cervical lymph nodes at presentation
* Distant metastatic disease (Stage IVC)
* Radiological evidence of gross extracapsular nodal tumor invasion
* Anatomy not allowing transoral access and exposure
* Prior head and neck cancer at any time (Other than BCC or SCC of skin)
* Coexistent second malignancy or history within 5 years of prior malignancy (other than BCC or early SCC skin or curatively treated Stage I carcinoma of cervix)
* Peripheral neuropathy >/= grade 1
* Have had prior Taxanes or Cisplatin
* Concurrent infection
* Coexisting medical illness of a severity that might interfere with treatment or follow-up, or who do not have the ability to give informed consent.
* Receiving any other investigational agent while on the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-08-14 (Actual); Primary Completion 2024-08-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Primary outcome: progression free survival. | 2 years
  Subjects will be evaluated for cancer recurrence or persistence. Index cancer recurrence or persistence following completion of treatment at any site will be recorded as an event. Progression free survival will be calculated at 2 years according to the Kaplan Meier methods.

SECONDARY OUTCOMES:
Disease Specific Survival (DSS) | 5 years
  The trial subjects will be followed for vital statistics (dead or alive) from the time enrolled in the trial. Any deaths that is caused by the index cancer will count as an event. DSS will be calculated with intention to treat analysis according to the Kaplan Meier methods at 5 years.
Overall Survival (OS) | 5 years
  The trial subjects will be followed for vital statistics (dead or alive) from the time of enrolment. Death from any cause will be counted as an event. Overall survival will be calculated according to the Kaplan Meier methods at years.
General Quality of Life (QOL) | 12 months.
  Patient-reported general quality of life outcome will be measured according to The European Organization for Research and Treatment of Cancer (EORTC) general quality of life questionnaire (EORTC QLQ-C30) at 3 month, 6 months, and 12 months following the completion of treatment. These questionnaires are validated and an integrated system for assessing the quality of life (QoL) of cancer patients participating in clinical trials. Outcome score for functional scales at 12 months will be compared to pretreatment levels.
Head and Neck Specific Quality of Life (QOL) | 12 months
  Patient-reported quality of life outcome will be measured according to EORTC head and neck specific questionnaire (QLQ-H&N35) prior to trial treatment (baseline), at 3 month, 6 months, and 12 months following the completion of treatment. These questionnaires are validated and an integrated system for assessing the quality of life (QoL) of head and neck cancer patients participating in clinical trials. Outcomes for symptom scales in H&N-35 at 12 months will be compared to pretreatment levels.

CONTACTS AND LOCATIONS:
Overall Officials: Nader Sadeghi, MD, Study Chair — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- McGill University Health Centre, Montreal, Quebec, Canada

REFERENCES:
- [Background] Sadeghi N, Mascarella MA, Khalife S, Ramanakumar AV, Richardson K, Joshi AS, Taheri R, Fuson A, Bouganim N, Siegel R. Neoadjuvant chemotherapy followed by surgery for HPV-associated locoregionally advanced oropharynx cancer. Head Neck. 2020 Aug;42(8):2145-2154. doi: 10.1002/hed.26147. Epub 2020 Mar 25. PMID 32212296
- [Background] Sadeghi N, Khalife S, Mascarella MA, Ramanakumar AV, Richardson K, Joshi AS, Bouganim N, Taheri R, Fuson A, Siegel R. Pathologic response to neoadjuvant chemotherapy in HPV-associated oropharynx cancer. Head Neck. 2020 Mar;42(3):417-425. doi: 10.1002/hed.26022. Epub 2019 Nov 27. PMID 31773857
- [Background] Sadeghi N, Li NW, Taheri MR, Easley S, Siegel RS. Neoadjuvant chemotherapy and transoral surgery as a definitive treatment for oropharyngeal cancer: A feasible novel approach. Head Neck. 2016 Dec;38(12):1837-1846. doi: 10.1002/hed.24526. Epub 2016 Jun 14. PMID 27299983